CLINICAL TRIAL: NCT04669925
Title: Tsunami Project - Description and Prediction of COVID-19 Impact on the Lombardy Region's Emergency System
Brief Title: COVID-19 Impact on the Lombardy Region's Emergency System
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: Tsunami
Record Dates: First submitted 2020-08-31; First posted 2020-12-17 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: Emergency Department; Emergency Medical Services
MeSH Terms: conditions — COVID-19; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Users of Lombardy Emergency System 2018-2020: Adults (affected or not affected by Covid-19) who asked for assistance to the Lombardy region's emergency system during the pandemic period and the previous two years

SUMMARY:
This study has 3 main goals:

* to quantitavely describe the Covid-19 impact on the organization and functioning of the Lombardy's emergency system;
* to create statistical model able to predict the flow of patients to the emergency room during the epidemic period and their destination (ex: discharge, hospitalization, death);
* to value the impact on the non Covid-19 patients, both for their possibility to receive medical treatment and as an outcome on their health

DETAILED DESCRIPTION:
The aim of this study is to evaluate the impact that Covid-19 had on the Emergency System of Lombardy. For instance, it affected the job organization and the possibility of responding to general health needs.

First of all, the study will consider the calls to the Emergency Medical Service, the number of accesses to the Emergency Department, the waiting time before hospitalization, the ED output home (discharge, hospitalization, death, self-discharge before the end of the visit).

Secondly, a statistical model will be implemented, in order to predict the number of patients in need of hospitalization for each day during the pandemic period. This model could help the re-organization of the hospital itself in case of a new Covid-19 outbreak.

Finally, it will evaluate the impact on non-Covid patients, to see the difference in the mortality trends and their possiblity to be cured in a proper way.

ELIGIBILITY:
Inclusion Criteria:

* over 18y

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who asked for assistance to the Lombardy region's emergency system during the pandemic period and the previous two years
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Daily calls to the Emergency System | jan 2020 - dec 2020
  The number of calls to the Lombardy Emergency System will be evaluated daily during the study period
Daily count of Emergency Department visits | jan 2020 - dec 2020
  The number of people accessing to each ED will be evaluated daily
Daily average boarding time | jan 2020 - dec 2020
  The average time between the end of the ED visit and the hospital admission will be measured daily
Outcome at ED discharge | jan 2020 - dec 2020
  Distribution of the ED outcome (home discharge, hospitalization, death, self-discharge before the end of the visit)
Mortality | jan 2020 - dec 2020
  Daily mortality for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (4):
- Italy (4):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Presidio Ospedaliero di Lodi, Lodi
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Carlo Borromeo, Milan

IPD SHARING:
Plan to Share IPD: Undecided
Protecting the privacy policy, all the data that underlie results in a publication will be shared. The scientific commettee of the study has to decide the criteria and the best way to share them